CLINICAL TRIAL: NCT03506022
Title: Prevalence of Sleep Apnea Syndrome in Patients With Type 1 Diabetes (APT1)
Brief Title: Prevalence of Sleep Apnea Syndrome in Patients With Type 1 Diabetes
Acronym: APT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2017_843_0019
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Sleep apnea syndrome, polysomnography and glucose monitoring continu glycemia (CGMS )
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: All patients over 18 years with type 1 mellitus diabetes will be included. The exclusion criteria are type-free diabetes (type 1 slow), age <18 years, a poor compliance with the follow-up (meetings unfulfilled without justification). All patients with known sleep disorders (OSA, narcolepsy, idiopathic hypersomnia).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with type 1 mellitus diabetes (Other): All participants were admitted in sleep laboratory and screened for one night of 8 hours employing standard polysomnography (Brainnet System - Medatec) parameters
  Interventions: Other: standard polysomnography

INTERVENTIONS:
Other: standard polysomnography — All participants were admitted in sleep laboratory and screened for one night of 8 hours employing standard polysomnography (Brainnet System - Medatec) parameters : electroencephalogram, electro-oculogram, electromyogram [chin], continuous nasal airflow body position, thoracic and abdominal strain gauges, haemoglobin oxygen saturation (SaO2) with an oximeter (Medatec) attached to finger. Blood pressure was measured in the evening during the physical examines, and then the CGMS recording startedpressure was measured in the evening during the physical examines, and then the CGMS recording started

SUMMARY:
Obstructive sleep apnea (OSA) and Type 2 diabetes are two frequent diseases that occur in adult population. The prevalence of OSA is higher in people with Type 2 diabetes compared with the general population7 ; in addition, the OSA syndrome is almost assessed in obese type 2 diabetes. The relationship between OSA and Type 2 diabetes has been well characterized: the OSA can contribute to increased insulin resistance or glucose intolerance; and, diabetes may worsen sleep-disordered breathing because of autonomic neuropathy8,9. The main link between OSA and Type 2 diabetes is central obesity, which triggers glucose intolerance/insulin resistance and is also an independent risk factor for OSA. Type 1 diabetes is generally not related to obesity; however, sleep-disordered breathing in these patients was described in few reports early as 1985 by pioneers such as Guilleminault5 and the prevalence of OSA is estimated at range 10 to 40% in type 1 diabetes patients. Few studies had evaluated the prevalence of sleep disorders in particular the sleep apnea syndrome in patients with type 1 diabetes and even less their influence on the glycemic control.

This study will take place at the CHU of Amiens-Picardie during a one-night hospitalization. The investigators will study in 44 type 1 diabetes mellitus (IAH apnea hypopnea index ≥15) who underwent polysomnography and continuous glucose monitoring of blood glucose

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years
* with type 1 mellitus diabetes

Exclusion Criteria:

* Type-free diabetes (type 1 slow),
* Age <18 years
* A poor compliance with the follow-up (meetings unfulfilled without justification).
* All patients with known sleep disorders (OSA, narcolepsy, idiopathic hypersomnia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of obstructive sleep apnea syndrome confirmed by polysomnography an apnea hypopnea Index ≥ 15 | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Amiens Picardie, Amiens, Picardie, France